CLINICAL TRIAL: NCT07053449
Title: The Impact of Treatment for Chronic Hepatitis B Virus on Non-clinical (Social) Harms Amongst Migrant Populations: A Qualitative Study. (B-SOCIAL)
Brief Title: The Impact of Treatment for Chronic Hepatitis B Virus on Non-clinical Harms
Acronym: B-SOCIAL
Status: Not yet recruiting | Type: Observational
Sponsor: Nottingham University Hospitals NHS Trust (Other)
Responsible Party: Sponsor
Other Study IDs: 24HP005
Record Dates: First submitted 2025-04-15; First posted 2025-07-08 (Actual); Last update posted 2025-07-16 (Actual); Status verified 2025-06

CONDITIONS: Hepatitis B Virus (HBV)
Keywords: Hepatitis B Virus; Qualitative; Lived Experience; Stigma
MeSH Terms: conditions — Hepatitis B; Social Stigma

STUDY DESIGN:
Observational Model: Other | Time Perspective: Other
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

GROUPS / COHORTS (1):
- HBsAg positive: Adult migrant populations living with chronic hepatitis B virus

SUMMARY:
The goal of this qualitative study is to explore the impact of antiviral treatment, or none, for chronic hepatitis B virus on the non-clinical (social) harms experienced by migrant populations living in the UK.

Two groups of participants living with hepatitis B virus will be interviewed, those taking the daily treatment, and those not prescribed any treatment.

DETAILED DESCRIPTION:
1. BACKGROUND Globally, chronic hepatitis B virus infection (HBV) is the most commonly occurring blood borne virus with approximately 300 million people infected. Infection with HBV can lead to the development of cirrhosis, resulting in liver failure or hepatocellular carcinoma (HCC). This is an important cause of preventable deaths, hence the World Health Organisation (WHO) objective to eliminate viral hepatitis as a public health problem by 2030. The WHO reported that globally, yearly deaths from acute and chronic viral hepatitis were approximately 1.4million, with 47% caused by HBV. Chronic HBV related global mortality in 2019 was estimated to be 331,000 attributable to cirrhosis, and 192,000 from hepatocellular cancer, all of which is entirely preventable if sufficient vaccination programmes were implemented for at-risk populations. The prevalence of HBV in England is estimated to be 268,767 (95% CI: 227,896 to 314,004), which equates to a prevalence of 0.58% (95% CI: 0.50% to 0.68%). HBV disproportionally affects people from global majority migrant populations who have relocated from lower income countries where prevalence rates are higher, largely Africa, South and South East Asia, and to a lesser extent Eastern Europe, predominantly due to mother to baby transmission and insufficient access to birth-dose preventative vaccines, iatrogenic transmission, and poor access to healthcare services. In the absence of antiviral treatment, the 5-year cumulative incidence of cirrhosis attributable to chronic HBV is between 8% and 20%. Finally, liver disease attributable to HBV is one cause of the inequalities in health outcomes experienced by ethnic populations that the NHS Race and Health Observatory are seeking to dissolve.

   There are a number of challenges when providing care to people with HBV infection. There are no symptoms until any resultant liver disease is advanced, the tests to diagnose and monitor it are complex and confusing to many healthcare professionals as well as patients and carers. Furthermore, HBV is most prevalent in populations at considerable social disadvantage, and it is associated with considerable stigmatization. The current oral treatments are also life-long. Treatment for HBV is currently initiated according to the physical factors that indicate the person is at increased risk of developing cirrhosis or acute liver failure, namely serum levels of HBV deoxyribonucleic acid (DNA), alanine transaminase (ALT), Hepatitis B e antigen (HBeAg) status, and the presence of liver fibrosis or cirrhosis, age, family history of hepatocellular carcinoma, or receiving immunosuppressant medication. There is a caveat in UK and European guidelines explaining that treatment may be offered for extra hepatic manifestations, but these refer to physical disorders such as vasculitis or glomerulonephritis rather than any non-clinical (social, cultural or psychological) manifestations. A report by the World Health Organisation (WHO) recommends an expansion to the criteria for treatment to reduce physical morbidity and mortality, but there is a current absence of data that explains the impact of treatment on the social domains of health.
2. RATIONALE The WHO however define health as being "…a state of complete physical, mental and social well-being and not merely the absence of disease and infirmity". Furthermore, holistic approaches to care view the person as a whole being and consider their social, psychological, and spiritual needs in addition to their physical health needs. The impact of living with chronic HBV infection in countries with a high prevalence has been shown to result in significant social harm, such as difficulty gaining employment, financial distress, and relationship difficulties. The holistic approach is at odds with the current biomedical model approach that focuses on the reduction of liver disease as the criteria for determining if and when to commence antiviral therapy for HBV. Whilst it is clear that the impact of living with HBV is more than the sum of the actual and potential physical ill-health, the specific role that treatments may have on the non-clinical, specifically social, outcomes has not been specifically unpacked. It is not clear for example, if treatment that leads to an undetectable viral load, considered to be a functional cure, reduces patient's experiences of felt or enacted stigma, social exclusion or relationship rejection.

A new HBV patient and public involvement and engagement group (PPIE) to identify research questions and advise on elements of study design has been created as part of an NIHR funded liver partnership, of which the chief investigator of this planned study is a member. An in-person meeting was held on 29.01.24 where individuals living with HBV and the British Liver Trust charity representatives remarked that patient-centred and holistic care had lost its meaning, and that most clinicians focused too heavily on the physical aspects of health. The PPIE group members agreed that a qualitative study to understand the role of antiviral therapy in mitigating against the social harms experienced by this population was a research priority.

Against this background, the aim of this qualitative study is to explore the impact of antiviral treatment, or none, for chronic HBV on the non-clinical (social) harms experienced by migrant populations living in the UK. Data will be obtained via semi-structured one to one interviews.

ELIGIBILITY:
Inclusion Criteria:

* Chronic HBsAg
* Able to give informed consent in English
* Able to converse in English
* Any migrant population member (non-UK) including if born overseas or in the UK
* Aged 18 years and over
* Has never taken antiviral treatment for HBV (12-15 participants)
* Prescribed and taking any oral treatment for HBV for a minimum of 12 months (12-15 participants)

Exclusion Criteria:

* Emotionally distressed due to HBV diagnosis
* Current episode of decompensated cirrhosis
* Current diagnosis of hepatocellular carcinoma

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Adults living with chronic hepatitis B virus infection
Sampling Method: Non-Probability Sample
Enrollment: 30 (Estimated)
Dates: Start 2025-08 (Estimated); Primary Completion 2025-12 (Estimated); Study Completion 2026-03 (Estimated)

PRIMARY OUTCOMES:
The qualitative Interview Topic Guide Questionnaire will thematically measure patients' experience of treatment, or not having treatment, for chronic hepatitis B virus infection. | The outcome measure will be assessed and data collected for reporting on day 1
  A qualitative interview topic guide questionnaire on patient's experience of treatment, or no treatment, for hepatitis B virus infection. The coding scheme will be inductively derived by the study team and overarching themes that characterise patients' experiences will be determined.

CONTACTS AND LOCATIONS:
Overall Officials: Kathryn E Jack, PhD, Principal Investigator — NUH

IPD SHARING:
Plan to Share IPD: No
There is no clinical or research rationale to share data

REFERENCES:
- [Background] Hsu YC, Huang DQ, Nguyen MH. Global burden of hepatitis B virus: current status, missed opportunities and a call for action. Nat Rev Gastroenterol Hepatol. 2023 Aug;20(8):524-537. doi: 10.1038/s41575-023-00760-9. Epub 2023 Apr 6. PMID 37024566
- [Background] Guidelines for the prevention, diagnosis, care and treatment for people with chronic hepatitis B infection [Internet]. Geneva: World Health Organization; 2024 Mar. Available from http://www.ncbi.nlm.nih.gov/books/NBK614989/ PMID 40424433
- [Background] World Health Organisation. (2023) What is the WHO definition of health? Available at: Frequently asked questions (who.int)
- [Background] World Health Organisation. (2016) WHO: Viral Hepatitis 2016-2021. June. https://apps.who.int/iris/bitstream/handle/10665/246177/WHO-HIV-2016.06-eng.pdf;sequence=1
- [Background] Wallace J, Pitts M, Liu C, Lin V, Hajarizadeh B, Richmond J, Locarnini S. More than a virus: a qualitative study of the social implications of hepatitis B infection in China. Int J Equity Health. 2017 Aug 1;16(1):137. doi: 10.1186/s12939-017-0637-4. PMID 28764768
- [Background] UK Health Security Agency (2024) Hepatitis B in the UK-2024 report. online available at: https://www.gov.uk/government/publications/hepatitis-b-in-england/hepatitis-b-in-england-2024#tab1
- [Background] UK Health Security Agency (2023) Hepatitis B in the UK-2023 report. Online available at: Hepatitis B in England - 2023 report (publishing.service.gov.uk)
- [Background] Tomar M, Sharma T, Prasad M. Social challenges experienced by Hepatitis B patients: A mixed method study. J Family Med Prim Care. 2023 Apr;12(4):748-755. doi: 10.4103/jfmpc.jfmpc_1575_22. Epub 2023 Apr 17. PMID 37312795
- [Background] Sharma S, Carballo M, Feld JJ, Janssen HL. Immigration and viral hepatitis. J Hepatol. 2015 Aug;63(2):515-22. doi: 10.1016/j.jhep.2015.04.026. Epub 2015 May 8. PMID 25962882
- [Background] Robertson, R., Williams, E., Buck., D., Breckwoldt, J. (2021). Ethnic health inequalities and the NHS: Driving progress in a changing system. Available at: https://www.nhsrho.org/wp-content/uploads/2023/05/Ethnic-Health-Inequalities-Kings-Fund-Report.pdf
- [Background] Papathanassiou, I. et al. (2013). Holistic Nursing Care: Theories and Perspectives. American Journal of Nursing Science. Vol. 2, No. 1, 2013, pp. 1-5. doi: 10.11648/j.ajns.20130201.11
- [Background] Oka T, Enoki H, Tokimoto Y, Kawanishi T, Minami M, Okuizumi T, Katahira K. Employment-related difficulties and distressed living condition in patients with hepatitis B virus: A qualitative and quantitative study. BMC Public Health. 2017 Jun 12;17(1):568. doi: 10.1186/s12889-017-4416-3. PMID 28606133
- [Background] Hepatitis B (chronic): diagnosis and management. London: National Institute for Health and Care Excellence (NICE); 2017 Oct. Available from http://www.ncbi.nlm.nih.gov/books/NBK553697/ PMID 32068988
- [Background] Fattovich G. Natural history of hepatitis B. J Hepatol. 2003;39 Suppl 1:S50-8. doi: 10.1016/s0168-8278(03)00139-9. No abstract available. PMID 14708678
- [Background] European Association for the Study of the Liver. EASL 2017 Clinical Practice Guidelines on the management of hepatitis B virus infection. J Hepatol. 2017 Aug;67(2):370-398. doi: 10.1016/j.jhep.2017.03.021. Epub 2017 Apr 18. PMID 28427875
- [Background] Adekanle O, Komolafe AO, Olowookere SA, Ijarotimi O, Ndububa DA. Hepatitis B Infection: A Mixed Methods of Disclosure Pattern and Social Problems in the Nigerian Family. J Patient Exp. 2020 Apr;7(2):208-216. doi: 10.1177/2374373519827965. Epub 2019 Mar 7. PMID 32851142